CLINICAL TRIAL: NCT04212299
Title: A Pilot Clinical Trial to Assess the Effect of Transfemoral Socket Design on Hip Muscle Function
Brief Title: Transfemoral Socket Design and Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Andrew Sawers, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0725; W81XWH1910507 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-12-20; First posted 2019-12-26 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Amputation

STUDY DESIGN:
Intervention Model Description: Transfemoral amputees who historically have worn an ischial containment prosthetic socket will be assessed at baseline, fit with the intervention (a sub-ischial socket), and then tested at 8 and 42 weeks after intervention. All comparisons will be made back to baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Baseline ischial containment to subischial socket (Experimental)
  Interventions: Device: Northwestern University Flexible Sub-Ischial Suction Socket (NU-FlexSIS)

INTERVENTIONS:
Device: Northwestern University Flexible Sub-Ischial Suction Socket (NU-FlexSIS) — The sub-ischial socket includes a firm, compressive, preferably cylindrical, fabric-covered silicone liner, a flexible inner socket, and a shorter rigid outer socket. The socket has proximal trim lines that do not impinge on the pelvis; they terminate distal to the ischial tuberosity and greater trochanter. For the NU-FlexSIS Socket, passive suction suspension is achieved using a one way valve and a liner with an internal seal.
  Since the prosthetic socket is a custom-made device, it is considered Class I exempt by the Food and Drug Administration (FDA).

SUMMARY:
The objective of this pilot research project is to evaluate the effect of prosthetic socket design on amputated limb hip muscle strength and endurance in Service members, Veterans, and civilians who use above-the-knee prostheses. Traditional above-the-knee socket designs provide pelvic support that interferes with hip motion. They may also reduce the effort required from amputated limb hip muscles to stabilize the hip and amputated limb, risking further loss of muscle mass and strength beyond that due to amputation. Long-standing use of above-the-knee sockets with pelvic support may therefore intensify amputated limb muscle loss and weakness, leading to challenges with walking and balance, increasing the effort required to walk, and contributing to degenerative changes in the hips and knees. Alternative socket designs that lessen the loss of muscle mass and strength are therefore required.

The investigators have developed a new socket without pelvic support for above-the-knee prosthesis users called the Northwestern University Flexible Sub-Ischial Suction (NU-FlexSIS) Socket. This new socket design increases user comfort and is often preferred by users over sockets with pelvic support. This new socket does not lessen the mechanical function of the socket, or walking and balance performance. Our recent research suggests that walking with this new socket may also increase amputated limb hip muscle size. However, more research is needed to demonstrate that this new socket design improves amputated limb hip muscle strength and endurance, leading to better function.

A socket design that increases amputated limb hip muscle strength and endurance would provide a simple way to restore amputated limb hip muscle weakness in above-the-knee prosthesis users. Despite a considerable decrease in hip muscle size and strength due to amputation surgery, amputated limb hip muscles are expected to compensate for the loss of knee and ankle function by providing stability and propulsion during walking. Walking in the new socket design without pelvic support is expected to increase amputated limb hip muscle strength and endurance, providing an appealing alternative to traditional resistance training in order to retain hip muscle strength. Unlike traditional resistance training, using this new socket design would not require additional time or equipment, and may be effective just by walking in the home, community, or workplace. Due to existing infrastructure (e.g., ongoing clinical adoption of the NU-FlexSIS Socket, existing instructional materials and courses for fabrication and fitting of the NU-FlexSIS Socket, as well as a continuing partnership with Chicago's largest provider of prosthetic clinical care), the investigators anticipate being able to translate our research results to clinical practice by the end of the project period.

The investigators expect the results of the proposed pilot research project to directly and positively benefit the health and well-being of Service members, Veterans, and civilians who are above-the-knee prosthesis users. Benefits of increasing amputated limb hip muscle strength and endurance may include: i) improved control over the prosthesis, ii) better balance, iii) reduced effort to walk, and iv) protection against joint degeneration. For Service members these benefits could improve their performance on challenging and/or uneven ground, and increase the distance and speed they can walk or run. For Veterans, these benefits could lead to greater independence during activities of daily living, and fewer falls, reducing the physical and emotional burden on family members and caregivers.

ELIGIBILITY:
Inclusion Criteria: worn an ischial containment socket for ≥ 2 years, able to walk short distances (10 meters), ability to read, write, and speak English, ≥ 2 years using a liner-based suspension, and a residual limb length ≥ 5".

Exclusion Criteria: amputation of a second leg, contralateral complications (e.g., hip replacement), or other major neuromusculoskeletal or cardiovascular conditions (e.g., heart failure).

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Baseline in Ischial Containment Socket
Arm/Group | Baseline Ischial Containment to Subischial Socket
Started | 5
Completed | 5
Not Completed | 0
Period: 8-week Follow up in Sub-ischial Socket
Arm/Group | Baseline Ischial Containment to Subischial Socket
Started | 5
Completed | 5
Not Completed | 0
Period: 42-week Follow up in Sub-ischial Socket
Arm/Group | Baseline Ischial Containment to Subischial Socket
Started | 5
Completed | 4
Not Completed | 1
Not completed — Participant experienced a heart attack | 1

BASELINE CHARACTERISTICS:
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (21.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Body mass [Mean (Standard Deviation); unit: kg] | 78.8 (6.81)
Height [Mean (Standard Deviation); unit: meters] | 1.73 (0.06)
Residual limb length [Mean (Standard Deviation); unit: cm] | 26 (3.2)
Time since amputation [Mean (Standard Deviation); unit: years] | 8 (7.5)
Cause of amputation [Count of Participants; unit: Participants]
  Traumatic | 3
  Dysvascular | 2
Medicare Functional Classification Level (K-Level) [Count of Participants; unit: Participants] — The Medicare Functional Classification Level (MFCL) K level is a 0 to 4 point scale of mobility for those with limb loss. A higher K level implies greater mobility potential. K-level determined by prosthetist.
  The MFCL levels are described as:
  K0 - Does not have the ability or potential to ambulate or transfer safely with a prosthesis K1 - Limited and unlimited household ambulator K2 - Limited community ambulator K3 - Community ambulator who has the ability to traverse most environmental barriers K4 - Potential for prosthetic ambulation that exceeds the basic ambulation skills
  Participants
    MFCL 1 | 0
    MFCL 2 | 1
    MFCL 3 | 4
    MFCL 4 | 0
Number of falls in past 12 months [Mean (Standard Deviation); unit: falls] | 2 (0.22)
Activities-specific Balance Confidence Scale score [Mean (Standard Deviation); unit: units on a scale 0 to 4] — Scale name: Activities-specific Balance Confidence (ABC) Scale
  Scale construct: balance self-efficacy
  Scale range (min/max): min = 0, max=4
  A higher ABC scale score implies greater balance self-efficacy (i.e., confidence)
  units on a scale 0 to 4 | 2.33 (0.32)
Prosthesis Limb Users Survey of Mobility [Mean (Standard Deviation); unit: units on a scale] — Scale name: Prosthetic Limb Users Survey of Mobility (PLUS-M) is a self-report instrument for measuring mobility of adults with lower limb amputation.
  Scale construct: perceived mobility
  Scale range (min/max): min = 21.8, max=71.4
  A higher PLUS-M score implies greater balance perceived mobility.
  units on a scale | 47.9 (1.81)

OUTCOME MEASURES:

1. Primary Outcome: Residual Limb Hip Muscle Peak Torque at Baseline
Description: Hip flexor, extensor, adductor and abductor muscle strength will be measured in transfemoral prosthesis users using a motor-driven isokinetic dynamometer. Muscular strength will be assessed via average peak torque (i.e., highest torque) across the first three repetitions of 12.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: newton-meters / kg*meters
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
newton-meters / kg*meters
  Hip extension | 25.6 [18.9 to 32.4]
  Hip flexion | 14.9 [7.29 to 22.6]
  Hip abduction | 25.6 [19.0 to 32.4]
  Hip adduction | 13.1 [8.63 to 17.5]

2. Primary Outcome: Residual Limb Hip Muscle Peak Torque at 8-weeks
Description: Hip flexor, extensor, adductor and abductor muscle strength will be measured in transfemoral prosthesis users using a motor-driven isokinetic dynamometer. Muscular strength will be assessed via average peak torque (i.e., highest torque) across the first three repetitions of 12. Comparison will be made to baseline measure.
Time Frame: 8 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: newton-meters / kg*meters
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
newton-meters / kg*meters
  Hip extension | 23.6 [15.2 to 31.9]
  Hip flexion | 14.1 [8.35 to 19.9]
  Hip abduction | 22.4 [15.4 to 29.5]
  Hip adduction | 13.3 [7.55 to 19.1]

3. Primary Outcome: Residual Limb Hip Muscle Peak Torque at 42-weeks
Description: as for outcome 2
Time Frame: 42 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: newton-meters / kg*meters
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
newton-meters / kg*meters
  Hip extension | 19.1 [9.12 to 29.1]
  Hip flexion | 12.2 [3.11 to 21.2]
  Hip abduction | 21.6 [8.77 to 34.4]
  Hip adduction | 10.1 [5.77 to 14.5]

4. Primary Outcome: Residual Limb Hip Muscle Endurance at Baseline
Description: Hip flexor, extensor, adductor and abductor muscle endurance will be measured in transfemoral prosthesis users using a motor-driven isokinetic dynamometer. Muscular endurance will be assessed via a fatigue index, calculated as a percentage of the difference between total work performed during the first and last 3 repetitions divided by total work over the first 3 repetitions. A higher fatigue index will be taken as evidence of reduced muscular endurance.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: newton-meters / kg*meters
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
newton-meters / kg*meters | NA [NA to NA] — Data were collected but could not be analyzed or summarized because most of the participants held back effort (i.e., self-paced) preventing an assessment of muscle endurance (i.e., change in peak torque from the first to the last trial). From this pilot protocol we have learned that in the future we need to use a single 30 second trial and look at changes from the first 3 seconds to the last 3 seconds for assessing hip muscle endurance in transfemoral prosthesis users.

5. Primary Outcome: Residual Limb Hip Muscle Endurance at 8-weeks
Description: Hip flexor, extensor, adductor and abductor muscle endurance will be measured in transfemoral prosthesis users using a motor-driven isokinetic dynamometer. Muscular endurance will be assessed via a fatigue index, calculated as a percentage of the difference between total work performed during the first and last 3 repetitions divided by total work over the first 3 repetitions. A higher fatigue index will be taken as evidence of reduced muscular endurance. Comparison will be made to baseline measure.
Time Frame: 8 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: newton-meters / kg*meters
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
newton-meters / kg*meters | NA [NA to NA] — Data were collected but could not be analyzed or summarized because most of the participants held back effort (i.e., self-paced) preventing an assessment of muscle endurance (i.e., change in peak torque from the first to the last trial). From this pilot protocol we have learned that in the future we need to use a single 30 second trial and look at changes from the first 3 seconds to the last 3 seconds for assessing hip muscle endurance in transfemoral prosthesis users.

6. Primary Outcome: Residual Limb Hip Muscle Endurance at 42-weeks
Description: as for outcome 5
Time Frame: 42 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: newton-meters / kg*meters
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
newton-meters / kg*meters | NA [NA to NA] — Data were collected but could not be analyzed or summarized because most of the participants held back effort (i.e., self-paced) preventing an assessment of muscle endurance (i.e., change in peak torque from the first to the last trial). From this pilot protocol we have learned that in the future we need to use a single 30 second trial and look at changes from the first 3 seconds to the last 3 seconds for assessing hip muscle endurance in transfemoral prosthesis users.

7. Primary Outcome: Residual Limb Hip Muscle Duration at Baseline
Description: Electromyographic (EMG) signals were recorded from transfemoral prosthesis users' residual limb muscles while walking. The duration of time each hip muscle was active during a stride was calculated as the percentage of the gait cycle (i.e., heel-strike to heel-strike) for which that EMG signal was above a baseline value (min: 0%, max: 100%). The larger the percentage of the gait cycle that a muscle was deemed to be active, the greater its duration.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
percentage
  Gluteus Maximus | 71.9 [52.1 to 91.6]
  Hamstrings | 73.2 [42.0 to 100.0]
  Gluteus medius | 76.5 [51.9 to 100.0]
  Tensor fascia latae | 78.7 [62.2 to 95.2]
  Rectus femoris | 81.3 [52.9 to 100.0]
  Adductor Magnus | 72.3 [52.3 to 92.4]

8. Primary Outcome: Residual Limb Hip Muscle Duration at 8-weeks
Description: as for outcome 7
Time Frame: 8 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
percentage
  Gluteus maximus | 64.0 [43.4 to 84.6]
  Hamstrings | 60.7 [26.6 to 94.8]
  Gluteus medius | 62.1 [22.5 to 100.0]
  Tensor fascia latae | 54.0 [33.0 to 75.0]
  Rectus femoris | 75.5 [49.7 to 100.0]
  Adductor magnus | 68.6 [32.1 to 100.0]

9. Primary Outcome: Residual Limb Hip Muscle Duration at at 42-weeks
Description: as for outcome 7
Time Frame: 42 weeks
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
percentage
  Gluteus maximus | 60.1 [29.8 to 90.3]
  Hamstrings | 61.1 [16.4 to 100.0]
  Gluteus medius | 51.3 [7.96 to 94.6]
  Tensor fascia latae | 45.1 [30.1 to 60.1]
  Rectus femoris | 75.9 [45.5 to 100.0]
  Adductor magnus | 53.0 [11.3 to 94.6]

10. Primary Outcome: Residual Limb Hip Muscle Integrated Area at Baseline
Description: Electromyographic (EMG) signals were recorded from transfemoral prosthesis users' residual limb muscles while walking. The total amount of hip muscle activity was calculated as the integrated area under the EMG signal during a gait cycle (i.e., heel-strike to heel-strike). Each EMG signal was normalized (i.e., divided by its maximum value across all the gait cycles and multiple by 100. The integrated areas is therefore reported as a percentage of that maximum (min: 0%, max: 100%). The larger the integrated area the more the muscle was deemed to be active.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: percentage of maximum value
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
percentage of maximum value
  Gluteus maximus | 23.4 [19.0 to 27.8]
  Hamstrings | 23.6 [8.71 to 38.5]
  Gluteus medius | 24.3 [12.5 to 36.2]
  Tensor fascia latae | 24.0 [17.9 to 29.9]
  Rectus femoris | 27.4 [16.3 to 38.6]
  Adductor magnus | 20.5 [13.7 to 27.4]

11. Primary Outcome: Residual Limb Hip Muscle Integrated Area at 8-weeks
Description: as for outcome 10
Time Frame: 8 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: percentage of maximum
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
percentage of maximum
  Gluteus maximus | 15.3 [3.53 to 27.1]
  Hamstrings | 14.4 [1.88 to 27.0]
  Gluteus medius | 28.0 [1.18 to 64.2]
  Tensor fascia latae | 13.4 [1.39 to 25.5]
  Rectus femoris | 24.2 [8.42 to 39.9]
  Adductor magnus | 22.7 [2.28 to 45.8]

12. Primary Outcome: Residual Limb Hip Muscle Integrated Area at 42-weeks
Description: as for outcome 10
Time Frame: 42 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: percentage of maximum
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
percentage of maximum
  Gluteus maximus | 30.9 [1.82 to 76.6]
  Hamstrings | 21.7 [1.99 to 46.5]
  Gluteus medius | 17.3 [1.10 to 40.6]
  Tensor fascia latae | 7.66 [2.94 to 12.38]
  Rectus femoris | 25.1 [5.69 to 44.6]
  Adductor magnus | 15.2 [2.37 to 39.7]

13. Primary Outcome: Peak Residual Limb Hip Muscle Activity at Baseline
Description: Electromyographic (EMG) signals were recorded from transfemoral prosthesis users' residual limb muscles while walking. The highest level of hip muscle activity was calculated as the peak of the EMG signal during a gait cycle (i.e., heel-strike to heel-strike). Each EMG signal was normalized (i.e., divided by its maximum value across all the gait cycles recorded during baseline). The peak EMG is therefore typically reported as a value between 0 and 1. However, if the peak value during assessments increases relative to baseline, the value of the peak activity will exceed 1. The larger the peak value the greater the activation of that muscle.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: mV
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
mV
  Gluteus maximus | 1.00 [NA to NA] — Peak muscle activity is amplitude normalized to its maximum value at baseline. Consequently all participants have a value of 1.0, creating no dispersion.
  Hamstrings | 1.00 [NA to NA] — Peak muscle activity is amplitude normalized to its maximum value at baseline. Consequently all participants have a value of 1.0, creating no dispersion.
  Gluteus medius | 1.00 [NA to NA] — Peak muscle activity is amplitude normalized to its maximum value at baseline. Consequently all participants have a value of 1.0, creating no dispersion.
  Tensor fascia latae | 1.00 [NA to NA] — Peak muscle activity is amplitude normalized to its maximum value at baseline. Consequently all participants have a value of 1.0, creating no dispersion.
  Rectus femoris | 1.00 [NA to NA] — Peak muscle activity is amplitude normalized to its maximum value at baseline. Consequently all participants have a value of 1.0, creating no dispersion.
  Adductor magnus | 1.00 [NA to NA] — Peak muscle activity is amplitude normalized to its maximum value at baseline. Consequently all participants have a value of 1.0, creating no dispersion.

14. Primary Outcome: Peak Residual Limb Hip Muscle Activity at 8 Weeks
Description: as for outcome 13
Time Frame: 8 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: mV
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
mV
  Gluteus maximus | 0.51 [0.23 to 0.78]
  Hamstrings | 0.71 [0.37 to 1.04]
  Gluteus medius | 1.46 [0.38 to 3.30]
  Tensor fascia latae | 0.71 [0.37 to 1.05]
  Rectus femoris | 0.82 [0.50 to 1.14]
  Adductor magnus | 0.90 [0.42 to 1.37]

15. Primary Outcome: Peak Residual Limb Hip Muscle Activity at 42 Weeks
Description: as for outcome 13
Time Frame: 42 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: mV
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
mV
  Gluteus maximus | 1.33 [0.09 to 2.57]
  Hamstrings | 0.85 [0.29 to 1.41]
  Gluteus medius | 1.29 [0.42 to 3.00]
  Tensor fascia latae | 0.47 [0.12 to 0.82]
  Rectus femoris | 1.18 [0.50 to 1.86]
  Adductor magnus | 0.65 [0.12 to 1.17]

16. Secondary Outcome: Four Square Step Test at Baseline
Description: A test of dynamic balance and coordination that assesses the participant's ability to step over objects forward, sideways, and backwards. Test was administered and scored as the best time (i.e., fastest) of two trials.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
seconds | 17.91 [6.63 to 29.2]

17. Secondary Outcome: Four Square Step Test at 8 Weeks
Description: as for outcome 16
Time Frame: 8-weeks after intervention
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
seconds | 15.1 [5.45 to 24.8]

18. Secondary Outcome: Four Square Step Test at 42 Weeks
Description: as for outcome 16
Time Frame: 42-weeks after intervention
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
seconds | 11.4 [7.13 to 15.7]

19. Secondary Outcome: One Leg Stance Test at Baseline
Description: A test of static balance that assesses the participant's ability to remain upright on one leg. Test was administered and scored as the best time (i.e., longest) of two trials. Longer times imply better static balance.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
seconds | NA [NA to NA] — Transfemoral prosthesis users were unable to stand on one leg at all, therefore the test was not performed.

20. Secondary Outcome: One Leg Stance Test at 8 Weeks
Description: as for outcome 19
Time Frame: 8 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
seconds | NA [NA to NA] — Transfemoral prosthesis users were unable to stand on one leg at all, therefore the test was not performed.

21. Secondary Outcome: One Leg Stance Test at 42 Weeks
Description: as for outcome 19
Time Frame: 42 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
seconds | NA [NA to NA] — Transfemoral prosthesis users were unable to stand on one leg at all, therefore the test was not performed.

22. Secondary Outcome: 10-Meter Walk Test at Baseline
Description: The 10MWT assesses walking speed in meters per second over a short duration. A faster speed is consider better walking performance. The fastest of 2 trials was used.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: meters/second
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
meters/second | 0.91 [0.57 to 1.24]

23. Secondary Outcome: 10-Meter Walk Test at 8 Weeks
Description: as for outcome 22
Time Frame: 8 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: meters/second
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
meters/second | 1.09 [0.78 to 1.40]

24. Secondary Outcome: 10-Meter Walk Test at 42 Weeks
Description: as for outcome 22
Time Frame: 42 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: meters/second
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
meters/second | 1.13 [0.89 to 1.36]

25. Secondary Outcome: 2-Minute Walk Test at Baseline
Description: The 2-Minute Walk Test is a measurement of waking endurance that assesses walking distance over two minutes. A longer distance walked indicates greater walking endurance.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
meters | 119 [71.1 to 167]

26. Secondary Outcome: 2-Minute Walk Test at 8 Weeks
Description: as for outcome 25
Time Frame: 8-weeks after intervention.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
meters | 122 [61.6 to 182]

27. Secondary Outcome: 2-Minute Walk Test at 42 Weeks
Description: as for outcome 25
Time Frame: 42-weeks after intervention.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
meters | 138 [93.3 to 182]

28. Secondary Outcome: Volume of Physical Activity at Baseline
Description: To assess the volume of physical activity, transfemoral prosthesis users wore a StepWatch4 activity monitor (Modus Health, Edmonds, WA) for a 2-week period. Activity bouts, or periods of time in which steps occur in successive 10-second intervals, will be derived from the step count data. The volume of physical activity will be quantified by the mean number of steps per activity bout. Higher values will be taken as evidence of greater physical activity.
Time Frame: 2 weeks prior to intervention (baseline)
Measure: Mean (95% Confidence Interval); unit: mean number of steps per activity bout
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
mean number of steps per activity bout | 27 [19 to 35]

29. Secondary Outcome: Volume of Physical Activity at 8 Weeks
Description: as for outcome 28
Time Frame: 8-weeks after intervention
Measure: Mean (95% Confidence Interval); unit: mean number of steps per activity bout
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
mean number of steps per activity bout | 30 [20 to 40]

30. Secondary Outcome: Volume of Physical Activity at 42 Weeks
Description: as for outcome 28
Time Frame: 42-weeks after intervention
Measure: Mean (95% Confidence Interval); unit: mean number of steps per activity bout
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
mean number of steps per activity bout | 34 [19 to 48]

31. Secondary Outcome: Frequency of Physical Activity at Baseline
Description: To assess the frequency of physical activity, transfemoral prosthesis users will wear a StepWatch4 activity monitor (Modus Health, Edmonds, WA) for a 2-week period. Activity bouts, or periods of time in which steps occur in successive 10-second intervals, will be derived from step count data. The frequency of physical activity will be quantified by the mean number of activity bouts per day. Higher values will be taken as evidence of greater physical activity.
Time Frame: 2 weeks prior to intervention (baseline)
Measure: Mean (95% Confidence Interval); unit: mean number of activity bouts per day
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
mean number of activity bouts per day | 63 [48 to 78]

32. Secondary Outcome: Frequency of Physical Activity at 8 Weeks
Description: as for outcome 31
Time Frame: 8 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: mean number of activity bouts per day
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
mean number of activity bouts per day | 74 [62 to 86]

33. Secondary Outcome: Frequency of Physical Activity at 42 Weeks
Description: as for outcome 31
Time Frame: 42 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: mean number of activity bouts per day
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
mean number of activity bouts per day | 81 [68 to 93]

34. Secondary Outcome: Duration of Physical Activity at Baseline
Description: To assess the duration of physical activity, transfemoral prosthesis users will wear a StepWatch4 activity monitor (Modus Health, Edmonds, WA) for a 2-week period. Activity bouts, or periods of time in which steps occur in successive 10-second intervals, will be derived from step count data. The duration of physical activity will be quantified by the mean time (in minutes) of activity bouts per day. Higher values will be taken as evidence of greater physical activity.
Time Frame: 2 weeks prior to intervention (baseline)
Measure: Mean (95% Confidence Interval); unit: mean time (in minutes) of activity bouts
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
mean time (in minutes) of activity bouts | 3.27 [2.87 to 3.67]

35. Secondary Outcome: Duration of Physical Activity at 8 Weeks
Description: as for outcome 34
Time Frame: 8 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: mean time (in minutes) of activity bouts
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 5
mean time (in minutes) of activity bouts | 3.68 [2.84 to 4.53]

36. Secondary Outcome: Duration of Physical Activity at 42 Weeks
Description: as for outcome 34
Time Frame: 42 weeks after intervention
Measure: Mean (95% Confidence Interval); unit: mean time (in minutes) of activity bouts
Arm/Group | Baseline Ischial Containment to Subischial Socket
Number analyzed (Participants) | 4
mean time (in minutes) of activity bouts | 3.76 [2.71 to 4.81]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 42 weeks.
Arm/Group | Baseline Ischial Containment to Subischial Socket
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
One participant dropped out prior to his week-42 follow up visit due to a medical condition unrelated to the study. Assessing hip muscle endurance as a decrease in performance over a set of 15 trials is not effective in transfemoral prosthesis users. Rather, a single 30 second trial, and comparing the first 3 and last 3 seconds is recommended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04212299/Prot_SAP_000.pdf